CLINICAL TRIAL: NCT01369550
Title: A Randomized, Controlled Trial to Assess the Effects of Stearidonic Acid-Containing Foods on Eicosapentaenoic Acid Levels of Red Blood Cells and the Omega-3 Index
Brief Title: Efficacy Study of Stearidonic Acid (SDA) Soybean Oil-containing Foods on Red Blood Cell Fatty Acid Content
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monsanto Company, LLC (Industry)
Collaborators: Solae, LLC (Industry)
Responsible Party: Shawna Lemke, Monsanto Company, LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PCR-10-263; PRV-10001 (Other: Provident Clinical Research & Consulting, Inc)
Record Dates: First submitted 2011-06-06; First posted 2011-06-09 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Healthy Volunteers; Markers of Cardiovascular Risk
MeSH Terms: interventions — Eicosapentaenoic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High-oleic sunflower oil-containing foods (Placebo Comparator): Subjects will consume 3 servings of foods containing high-oleic sunflower oil plus 3x500 mg high-oleic sunflower oils softgels per day.
  Interventions: Other: High-oleic sunflower oil containing foods
- Eicosapentaenoic acid (Active Comparator): Subjects will consume 3 x 500 mg eicosapentaenoic acid ethyl ester in softgels plus 3 servings of high-oleic sunflower oil-containing foods per day
  Interventions: Other: Eicosapentaenoic acid
- SDA soybean oil-containing foods (Experimental): Subjects in this arm will consume 3 servings of SDA soybean oil-containing foods plus 3 x 500 mg high-oleic sunflower oil softgels per day.
  Interventions: Other: SDA soybean oil-containing foods

INTERVENTIONS:
Other: SDA soybean oil-containing foods — 3 servings per day of foods containing 500 mg each SDA soybean oil plus 3 x 500 mg high-oleic sunflower oil in softgels per day.
  Arms: SDA soybean oil-containing foods
Other: High-oleic sunflower oil containing foods — 3 servings per day of foods containing 500 mg high-oleic sunflower oil plus 3 x 500 mg high-oleic sunflower oil in softgels per day
  Arms: High-oleic sunflower oil-containing foods
Other: Eicosapentaenoic acid — 3 x 500 mg per day of Eicosapentaenoic acid as an ethyl ester in softgels plus 3 servings per day of high-oleic sunflower oil-containing foods
  Arms: Eicosapentaenoic acid

SUMMARY:
The purpose of this clinical trial is to evaluate whether the omega-3 fatty acid stearidonic acid (SDA), when used as a food ingredient, increases the level of the long-chain omega-3 fatty acid eicosapentaenoic acid (EPA) in red blood cell (RBC) membranes in men and women.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female, 21 to 65 years of age, inclusive.
2. Body mass index (BMI) ≥18.00 and <40.00 kg/m2 at visit 1, week -2.
3. Subject has no health conditions that would prevent him/her from fulfilling the study requirements as judged by the Investigator on the basis of medical history and routine laboratory test results.
4. Subject is willing to avoid alcohol consumption for 24 h prior to every clinic visit.
5. Subject has no plans to change smoking habits during the study period.
6. Subject is willing to maintain a stable body weight, activity level and dietary pattern except for use of the study products, as directed.
7. Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

1. Subject has coronary heart disease or a coronary heart disease risk equivalent including any of the following:

   1. Diabetes mellitus (or fasting glucose ≥126 mg/dL at visit 1, week -2);
   2. Clinical signs of atherosclerosis including peripheral arterial disease, abdominal aortic aneurysm, carotid artery disease [symptomatic (e.g., transient ischemic attack or stroke of carotid origin) or >50% stenosis on angiography or ultrasound] or other forms of clinical atherosclerotic disease (e.g., renal artery disease);
   3. Presence of multiple risk factors that give a person a greater than 20% chance for developing coronary artery disease within 10 years. This will be determined by the Framingham risk index calculated at visit 1, week -2.
2. Abnormal laboratory test results of clinical significance, including, but not limited to creatinine ≥1.5 mg/dL and ALT or AST ≥1.5X the upper limit of normal at visit 1, week -2.
3. TG ≥400 mg/dL at visit 1, week -2.
4. Subject smokes more than one pack of cigarettes (20 cigarettes) per day.
5. Subject has a history or presence of clinically important renal, hepatic, pulmonary, biliary, gastrointestinal, neurologic or endocrine disorders that in the judgment of the Investigator, would interfere with the subject's ability to provide informed consent, comply with the study protocol (which might confound the interpretation of the study results), or put the subject at undue risk. Stable, treated hypothyroidism is allowed.
6. Uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg as defined by the average blood pressure measured at visit 1, week -2). One re-test will be allowed on a separate day prior to visit 2, week 0 for subjects whose blood pressure exceeds either of these cut points at visit 1, week -2.
7. Unstable use (initiation or change in dose) within four weeks of visit 1 (week -2; Appendix 1) of antihypertensive medications or thyroid hormone replacement.
8. Use of any lipid-altering drugs, including statins, bile acid sequestrants, cholesterol absorption inhibitors, fibrates, or prescription formulations of niacin within four weeks of visit 1 (week -2) and throughout the study. If a subject needs to wash off of a drug, he/she will be consented and then asked to return after the four week washout.
9. Use of EPA/DHA from a drug or supplement within four months of visit 1, week -2 and throughout the study period. If subject has used >1.0 g/d of EPA, DHA, or combination of EPA and DHA from a drug or supplement, use must have been discontinued at least six months prior to the visit 1, week -2 blood draw.
10. Frequent use (more than twice per month) of any non-study-related EPA/DHA containing enriched foods (such as DHA-enriched eggs) within four months of visit 1, week -2 and avoidance of these enriched foods throughout the study period.
11. Use of ALA-containing seeds and oils (i.e., flaxseed, perilla seed, hemp, spirulina, walnut, mustard seed or black currant oil) for more than one week duration within four weeks of visit 1, week -2 and throughout the study period.
12. Consumption of fatty fish (salmon, herring, mackerel, albacore tuna, or sardines) more than twice per month within four months of visit 1, week -2. Unwillingness to avoid all fish, except shellfish and crustaceans, throughout the study period (Appendix 6. Note: it is recognized that many fish are not significant sources of omega-3 fatty acids; however, these foods are restricted to simplify the dietary advice in this low-dose SDA study).
13. Use of any dietary supplement known to alter lipid metabolism, including but not limited to: dietary fiber supplements, red rice yeast supplements, garlic supplements, soy isoflavone supplements, sterol/stanol products, policosanols, niacin or its analogues at doses >50 mg/d, or others at the discretion of the Investigator within the four weeks prior to visit 1, week -2 or during the study. If a subject needs to discontinue a lipid-altering supplement(s), he/she will washout for four weeks prior to the screening visit procedures (visit 1, week -2).
14. Use of any weight-loss medication (prescription or over-the counter) including, but not limited to, lipase inhibitors [orlistat (alli™)], within four weeks prior to visit 1, week -2 and throughout the study.
15. Use of any weight loss supplement or program within four weeks of visit 1, week -2 and throughout the study.
16. Known allergy or sensitivity to study products or any ingredients of the study products (study products may contain milk, soy or wheat).
17. Subject has a history or presence of cancer in the prior two years, except for non-melanoma skin cancer (e.g., basal or squamous cell carcinoma of the skin).
18. Females who are pregnant, planning to be pregnant during the study period, lactating, or women of childbearing potential who are unwilling to commit to the use of a medically approved form of contraception throughout the study period. The method of contraception must be recorded in the source documentation.
19. Current or recent history of (within 12 months of visit 1, week -2) or strong potential for alcohol or substance abuse. Alcohol abuse will be defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1 ½ oz distilled spirits).
20. Exposure to any non-registered drug product within 30 days prior to the screening visit (visit 1, week -2).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
EPA as a percent of total of fatty acids in red blood cell membranes | 12 weeks
Omega-3 Index | 12 weeks
  Sum of EPA + DHA as a % of total fatty acids in the red blood cell membrane

SECONDARY OUTCOMES:
Fasting Triglycerides | 12 weeks
Fasting Insulin | 12 weeks
HOMA-IR | 12 weeks
  Homeostasis model assessment of insulin resistence
HOMA-%B | 12 weeks
  Homeostasis model assessment - Beta-cell function
SDA as a percent of total fatty acids in the red blood cell | 12 weeks
Docosapentaenoic acid (DPA) as a percent of total fatty acids in the red blood cell membrane | 12 weeks
Arachidonic acid (AA) as a percent of total fatty acids in red blood cell membranes | 12 weeks
Fasting serum chemistry | 12 weeks
  Standard panel containing: glucose, calcium, sodium, potassium, BUN, creatinine, ALP, ALT, AST, GGT, Total bilirubin, BUN:creatinine ratio, amylase, uric acid, CPK.
Fasting Hematology Profile | 12 weeks
  Standard panel containing: WBC count, WBC with differential, RBC count, hemoglobin, hematocrit,platelet count
Fasting lipid panel | 12 weeks
  Total cholesterol, LDL-C, HDL-C, non-HDL-C, TC/HDL-C

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Maki, PhD, Study Director — Provident Clinical Research & Consulting, Inc.
Locations (2):
- United States (2):
  - Meridien Research, St. Petersburg, Florida
  - Provident Clinical Research & Consulting, Inc., Addison, Illinois